CLINICAL TRIAL: NCT00364858
Title: A Phase IV, Multicenter, Randomized, Dose Frequency Study of the Safety and Efficacy of Cerezyme® Infusions Every Four Weeks Versus Every Two Weeks in the Maintenance Therapy of Patients With Type 1 Gaucher Disease
Brief Title: Safety and Efficacy of Cerezyme® Infusions Every 4 Weeks Versus Every 2 Weeks in Type 1 Gaucher Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZ-011-01
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Gaucher Disease, Type 1; Cerebroside Lipidosis Syndrome; Glucocerebrosidase Deficiency Disease; Glucosylceramide Beta-Glucosidase Deficiency Disease; Gaucher Disease, Non-Neuronopathic Form
Keywords: Type 1 Gaucher Disease; Glucocerebrosidase Deficiency Disease
MeSH Terms: conditions — Gaucher Disease | interventions — imiglucerase

ARMS (2):
- Q2 Cerezyme (Other): Patients receiving Cerezyme one infusion every 2 weeks (Q2).
  Interventions: Drug: Cerezyme
- Q4 Cerezyme (Other): Patients receiving Cerezyme one infusion every 4 weeks (Q4).
  Interventions: Drug: Cerezyme

INTERVENTIONS:
Drug: Cerezyme — Cerezyme doses of 20-60U/kg every 2 weeks (Q2 Arm) or 40-120 U/kg every 4 weeks (Q4 Arm).

SUMMARY:
This is a multicenter, randomized trial to compare the safety and efficacy of two dosing frequencies of Cerezyme® in patients with Gaucher disease who are currently being treated with Cerezyme®.

Approximately 90 patients will be randomized in a 2:1 (q4 : q2) ratio to one of two treatment arms at up to 26 study centers worldwide. Patients will continue to receive the same total 4-week dose that they were receiving prior to study enrollment, however, they will be randomized to receive either their total 4-week dose in two infusions, one infusion every 2 weeks or their total 4-week dose in one infusion every 4 weeks. The randomization scheme will ensure a 2:1 balance between the every 4-week versus every 2-week infusion groups, respectively.

ELIGIBILITY:
Inclusion Criteria:

* The patient must provide written informed consent prior to undergoing any study-related procedures.
* The patient has a confirmed diagnosis of Gaucher disease with a documented deficiency of glucocerebrosidase by enzyme assay
* The patient has been genotyped or will have genotyping performed within 3 months of study enrollment.
* The patient has been treated with Cerezyme for at least 2 years prior to study enrollment.
* The patient has been on a stable dose of between 20-60 U/kg every 2 weeks for at least 6 months prior to study enrollment.
* The patient is at least 18 years old.
* The patient has a hemoglobin value of ≥ 11.0 g/dL for women and ≥ 12.0 g/dL for men and a platelet count of ≥ 100,000 mm^3.
* The patient's liver volume is ≤ 1.8 x normal confirmed by MRI or CT within 6 months of randomization.
* The patient's spleen volume is ≤ 10 x normal confirmed by MRI or CT within 6 months of randomization.
* The patient has a serum creatinine < 2.0 mg/dL, an ASTand ALT < 2 x upper limit of normal and a total bilirubin < 2.0 x upper limit of normal.
* Female patients of childbearing potential must have a negative pregnancy test within 2 weeks prior to randomization into the study.

Exclusion Criteria:

* The patient is pregnant.
* The patient has evidence of neurologic or pulmonary involvement with Gaucher disease confirmed by medical history.
* The patient has evidence of current or prior bleeding varices or liver infarction requiring hospitalization confirmed by medical history.
* The patient has evidence of pathologic bone fractures, medullary infarctions, lytic lesions or avascular necrosis secondary to Gaucher disease confirmed by skeletal evaluation within 6 months of randomization.
* The patient has had a bone crisis (defined as pain with acute onset which requires immobilization of the affected area, narcotics for relief of pain and may be accompanied by periosteal elevation, increased white cell count, fever or debilitation of > 3 days) within 12 months of randomization.
* Patient has received an investigational drug within 30 days of the start of their participation in this trial. Patients may not receive any other investigational product throughout the course of the study.
* The patient has a clinically significant disease (with the exception of symptoms relating to Gaucher disease), including clinically significant cardiovascular, hepatic, immunologic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstances that, in the opinion of the Investigator, would preclude participation in the trial or potentially decrease survival
* Patient has a medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the patient's compliance with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2001-12; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kaye, M.D., Study Director — Genzyme, a Sanofi Company
Locations (26):
- United States (18):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University Research Foundation for Lysosomal Storage Disease, Inc., Coral Springs, Florida
  - Emory University, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Midwest Cancer Research Group, Inc., Skokie, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Institute for Genetics Medicine Saint Peter's University Hospital, New Brunswick, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Hemophilia Center of Western New York, Buffalo, New York
  - New York Oncology/Hematology PC, Latham, New York
  - New York University, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Research Foundation, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Estadual de Hematologia Arthur de Siqueira Cavalcanti (HEMORIO), Rio de Janeiro, Brazil
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Italy (3):
  - Istituto Giannina Gaslini, Genova
  - Universita degli Studi di Napoli "Federico II", Naples
  - Istituto per l'Infanzia Burlo-Garofolo, Trieste
- Instytut Pomnik Centrum Zdrowia Dzeicka, Warsaw, Poland
- Hospital Vall d´Hebrón, Barcelona, Spain
- Royal Free Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were randomized 2:1 to receive Cerezyme either once every 4 weeks (Q4) or once every 2 weeks (Q2) for 24 months. The studied period was from 14 December 2001 through 01 February 2007. There were 26 centers worldwide (18 United States, 1 Canada, 6 Europe, and 1 Brazil); 25 centers randomized patients to treatment.
Groups:
- Q4 Cerezyme: Patients receiving Cerezyme one infusion every 4 weeks(Q4).
Period: Overall Study
Arm/Group | Q2 Cerezyme | Q4 Cerezyme
Started | 33 | 62
Completed | 26 | 40
Not Completed | 7 | 22
Not completed — Adverse Event | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Clinical failure | 2 | 13
Not completed — Discontinuation at baseline | 1 | 0
Not completed — Non-compliant | 1 | 0
Not completed — Return to Q2 regimen | 0 | 1
Not completed — Clinical baseline issue | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Q2 Cerezyme | Q4 Cerezyme | Total
Number analyzed (Participants) | 33 | 62 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (17.40) | 47.8 (14.47) | 46.8 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 34 | 47
  Male | 20 | 28 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success at Month 24/Discontinuation
Description: Patients are considered to be a clinical success if ALL of the following are met: The patient's hemoglobin does not fall more than 1.25g/dL for women or 1.5 g/dL for men below the patient's baseline value, platelet count does not fall more than 25% below the patient's baseline value or does not fall below 80,000 mm3, liver and spleen volumes are not greater than 20% above the patient's baseline value, no evidence of bone disease progression, including no incidence of pathologic fractures, medullary infarctions, lytic lesions or avascular necrosis and has had no bone crises during the study.
Time Frame: Month 24 (or at time of discontinuation)
Population: Intent-to-Treat (ITT) Population. All patients who enrolled in the study and received AT LEAST ONE infusion were included in the ITT population.
Measure: Number; unit: patients
Arm/Group | Q2 Cerezyme | Q4 Cerezyme
Number analyzed (Participants) | 26 | 57
patients
  Number of participants with Clinical Success | 21 | 36
  Proportion of participants with Clinical Success | 0.808 | 0.632
Statistical Analysis 1: Comparison: Q2 Cerezyme vs Q4 Cerezyme; Difference in proportion of Clinical Success = (Proportion of participants with Clinical Success Q4 - Proportion of participants with Clinical Success Q2); Test type: Superiority or Other; Agresti and Min = -0.176, 95% CI [-0.357 to 0.058]

2. Secondary Outcome: Mean Composite Scores of the SF-36 Health Survey at Baseline
Description: The mean composite scores (0 being worst and 100 being best) for both treatment groups at Baseline. Composite scores for both treatment groups approximated those of the general population at baseline and at Month 24.
Time Frame: Baseline
Population: Quality of life was evaluated and measured by the SF-36 questionnaire.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Q2 Cerezyme | Q4 Cerezyme
Number analyzed (Participants) | 33 | 61
Units on a scale
  Composite Physical Health | 49.8 (8.41) | 46.9 (10.26)
  Composite Mental Health | 52.9 (7.6) | 53.0 (8.47)

3. Secondary Outcome: Mean Composite Scores of the SF-36 Health Survey at Month 24/Discontinuation.
Description: The mean composite scores (0 being worst and 100 being best) for both treatment groups at Month 24/Discontinuation. The mean composite scores for both treatment groups approximated those of the general population at baseline and at Month 24.
Time Frame: Month 24 (or at time of discontinuation)
Population: Quality of life was evaluated and measured by the SF-36 questionnaire.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Q2 Cerezyme | Q4 Cerezyme
Number analyzed (Participants) | 25 | 53
Units on a scale
  Composite Physical Health | 49.1 (7.52) | 46.2 (12.39)
  Composite Mental Health | 53.8 (8.47) | 52.6 (7.35)

4. Secondary Outcome: Mean Change From Baseline in Composite Scores of the SF-36 Health Survey at Month 24/Discontinuation
Description: The mean composite scores (0 being worst and 100 being best) for both treatment groups approximated those of the general population at baseline. Composite score - The overall composite scores were comprised of a standardized physical and mental component score.
Time Frame: Baseline and Month 24 (or at time of discontinuation)
Population: Quality of life was evaluated and measured by the SF-36 questionnaire.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Q2 Cerezyme | Q4 Cerezyme
Number analyzed (Participants) | 25 | 52
Units on a scale
  Composite Physical Health | -1.5 (7.40) | -0.5 (7.33)
  Composite Mental Health | 0.6 (6.48) | -0.5 (7.34)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Q2 Cerezyme | Q4 Cerezyme | Total
Serious Adverse Events (participants affected / at risk) | 7/33 | 4/62 | 11/95
Other Adverse Events (participants affected / at risk) | 20/33 | 51/62 | 71/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Q2 Cerezyme (N=33) | Q4 Cerezyme (N=62) | Total (N=95)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Blindness (Eye disorders) | 0 | 1 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Parkinson's disease (Nervous system disorders) | 2 | 0 | 2
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Aortic dilatation (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Q2 Cerezyme (N=33) | Q4 Cerezyme (N=62) | Total (N=95)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Cardiomegaly (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 | 1 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 2 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 2
Vision blurred (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 3
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 1 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Asthenia (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 0 | 6 | 6
Feeling hot (General disorders) | 0 | 1 | 1
Ill-defined disorder (General disorders) | 0 | 1 | 1
Infusion site erythema (General disorders) | 0 | 1 | 1
Infusion site pain (General disorders) | 0 | 2 | 2
Irritability (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 2 | 2
Pyrexia (General disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Multiple allergies (Immune system disorders) | 0 | 1 | 1
Acariasis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 3 | 3
Bronchitis acute (Infections and infestations) | 0 | 2 | 2
Cystitis (Infections and infestations) | 0 | 2 | 2
Furuncle (Infections and infestations) | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 4 | 4
Influenza (Infections and infestations) | 0 | 4 | 4
Laryngitis (Infections and infestations) | 1 | 1 | 2
Nail bed infection (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3 | 4
Otitis externa (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Sinusitis (Infections and infestations) | 2 | 5 | 7
Tinea versicolour (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1 | 2
Mountain sickness acute (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 2
Spinal cord injury lumbar (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Antibody test positive (Investigations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 1
Breath sounds abnormal (Investigations) | 1 | 0 | 1
Cardiac murmur (Investigations) | 0 | 1 | 1
Computerised tomogram abdomen abnormal (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 5 | 5
Platelet count decreased (Investigations) | 0 | 5 | 5
Prostatic specific antigen increased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 1 | 0 | 1
White blood cells urine positive (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 10 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 10 | 10
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervical root pain (Nervous system disorders) | 1 | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 3
Headache (Nervous system disorders) | 2 | 6 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Intention tremor (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0 | 1
Parkinsonian gait (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2 | 2
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1
Affect lability (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 2
Depression (Psychiatric disorders) | 1 | 1 | 2
Listless (Psychiatric disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia effluvium (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria localised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 3 | 4
Hypotension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.